CLINICAL TRIAL: NCT00051259
Title: A Multicenter, Double-Blind, Randomized, Placebo Controlled Comparison of the Effects on Sexual Functioning of Extended-Release Bupropion Hydrochloride (300-450mg) and Escitalopram (10-20mg) in Outpatients With Moderate to Severe Major Depression Over an Eight-Week Treatment Period
Brief Title: Effects of Antidepressants on Sexual Functioning
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK130926
Record Dates: First submitted 2003-01-07; First posted 2003-01-08 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: depression; MDD; sexual dysfunction; orgasm disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological

INTERVENTIONS:
Drug: Extended-Release Bupropion Hydrochloride

SUMMARY:
The purpose of this trial is to study the effects of two depression medications on sexual functioning.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Major Depressive Disorder (MDD) with current duration lasting 12 weeks but no greater than 2 years.
* Subjects must engage in sexual activity that leads to orgasm at least once every two weeks.
* Subject must have normal orgasmic function and be willing to discuss with investigator.

Exclusion Criteria:

* Subjects that have arousal or orgasm dysfunction.
* Has previously failed to respond to two adequate trials of antidepressants in past 2 years.
* Subject has other unstable medical disorders.
* Subject has a positive urine test for illicit drug use at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 2003-01; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with orgasm dysfunction. Change in HAMD-17 total score.

SECONDARY OUTCOMES:
Percent of subjects in remission, HAMD-17. Changes in Sexual Functioning Questionnaire. Percent of responders, HAMD-17 CGI-I and CGI-S.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (23):
- United States (23):
  - GSK Investigational Site, Berkeley, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Coral Springs, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Terre Haute, Indiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Lincoln, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Madison, Wisconsin